CLINICAL TRIAL: NCT01268046
Title: The Effect of Low Dose Estrogen on Cortical Function as a Function of Age in Postmenopausal Women.
Brief Title: Aging and Estrogen on Cortical Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Associate Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2009P-002311; R01AG013241 (NIH)
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Memory Loss; Cognitive Changes; Postmenopausal Symptoms
Keywords: aging; postmenopausal women; estrogen; memory
MeSH Terms: conditions — Memory Disorders | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Each participant was randomized to placebo or estrogen using a block randomized design by age group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization was performed by the Research Pharmacy and the investigative team was blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Young postmenopausal women - estrogen (Experimental): transdermal estrogen patch OR estradiol oral capsule for 1 month
  Interventions: Drug: Estradiol oral capsule; Drug: transderman estrogen patch
- Older postmenopausal women - estrogen (Experimental): transdermal estrogen patch OR estradiol oral capsule for 1 month
  Interventions: Drug: Estradiol oral capsule; Drug: transderman estrogen patch
- Young postmenopausal women - placebo (Placebo Comparator): transdermal placebo patch for 1 month or placebo oral capsule for 1 month
  Interventions: Drug: trasdermal placebo patch; Drug: placebo oral capsule
- Older postmenopausal women - placebo (Placebo Comparator): transdermal placebo patch for 1 month or placebo oral capsule for 1 month
  Interventions: Drug: trasdermal placebo patch; Drug: placebo oral capsule

INTERVENTIONS:
Drug: Estradiol oral capsule — 1 oral capsule (1 mg estradiol) administered daily for one month
  Other Names: Micronized Estradiol; Estradiol
  Arms: Older postmenopausal women - estrogen; Young postmenopausal women - estrogen
Drug: transderman estrogen patch — transdermal estrogen patch (50 mcg/day) for one month
  Other Names: Climara; Estraderm; Estrogen patch
  Arms: Older postmenopausal women - estrogen; Young postmenopausal women - estrogen
Drug: trasdermal placebo patch — transdermal placebo patch with patch change every 84 hr for one month
  Other Names: Placebo patch
  Arms: Older postmenopausal women - placebo; Young postmenopausal women - placebo
Drug: placebo oral capsule — placebo oral capsule administered daily for one month.
  Other Names: Placebo capsule
  Arms: Older postmenopausal women - placebo; Young postmenopausal women - placebo

SUMMARY:
This study will focus on how estrogen affects parts of the brain associated with memory and how the effect of estrogen is altered with aging in postmenopausal women.

DETAILED DESCRIPTION:
The broad goal of this proposal is to determine the effect of aging on areas of the brain whose function is impacted by gonadal steroids in women. The overarching hypothesis is that aging differentially alters the effects of estrogen on the brain. Our preliminary data indicated that aging alters the effect of estrogen on brain regions involved in cognition and thus, the current study focused on the impact of aging on functional changes induced by estrogen in cortical and subcortical areas associated with verbal working memory and declarative/episodic memory.

As our model, we will use women in whom the absence of gonadal function makes it possible to control the duration and amount of estrogen exposure, specifically postmenopausal women who are younger (45-55) or older (65-80) who receive either oral or transdermal estradiol to achieve premenopausal early follicular phase estradiol levels.. We evaluate the effects of low dose estrogen exposure at 48 hr and 1 month to determine whether the short-term changes in brain regions involved in cognition with low dose estrogen exposure seen in our preliminary studies are confirmed and whether changes with short-term estrogen exposure persist with more prolonged exposure, a finding that would have enormous clinical relevance. These studies, using sophisticated neuroimaging tools (structural and functional magnetic resonance imaging [MRI] and [18F] 2-fluoro-2-deoxy-D-glucose positron emission tomography [FDG-PET]), provide a unique window into the brain in women.

ELIGIBILITY:
Inclusion Criteria:

1. young postmenopausal (age 45-55) or older (age 65-80) postmenopausal women
2. otherwise healthy, non-obese women with normal blood pressure and a history of normal menopause, defined by the absence of menses for at least 12 months
3. prescription hormone replacement treatment discontinued at least 3 months before study
4. Normal or corrected normal vision
5. Intelligence quotient (IQ) > 70 on the Wechsler Adult Reading Test (WTAR)*
6. Absence of Mild Cognitive Impairment (MCI) and depression on the Mini Mental State Examination (MMSE)** and Beck Depression Inventory II (BDI-II).***
7. Normal mammogram or breast MRI within the past 2 years

Exclusion Criteria

1. On gonadal hormone replacement medication, herbal supplements and/or over the counter menopause treatment within three months of study
2. History of radiotherapy or chemotherapy.
3. Absolute contraindications to the use of physiologic replacement doses of estrogen and/or history of coronary artery disease
4. History of breast cancer, blood clot, pulmonary embolus, hypercoagulability and stroke.
5. On centrally acting medications
6. History of head trauma and/or neurologic disorder
7. Contraindication to MRI (eg. metal implants) or PET imaging (eg. PET imaging studies in the previous 12 months)
8. Concurrent participation in research studies involving medications and/or PET scans.
9. Left handedness.
10. Current breast lump(s) or family/genetic history of breast cancer in younger women (< 40 years old).
11. Current smoking

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Reproductive Endocrine Unit, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information will be made available on request to the PI once the primary data analysis has been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From time of publication of initial 2 manuscripts (December 2019) for 5 years
Access Criteria: Academic investigator with funding for analysis, approval of PI

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Postmenopausal Women - Estrogen: 1 oral capsule (1 mg estradiol) administered daily for one month OR 1 transdermal estrogen patch (50 mcg/day) with patch change every 84 hr for one month in younger postmenopausal women
- Older Postmenopausal Women - Estrogen: 1 oral capsule (1 mg estradiol) administered daily for one month OR 1 transdermal estrogen patch (50 mcg/day) with patch change every 84 hr for one month in older postmenopausal women
- Young Postmenopausal Women - Placebo: 1 placebo capsule administered daily for one month OR 1 placebo patch with patch change every 84 hr for one month in younger postmenopausal women
- Older Postmenopausal Women - Placebo: 1 placebo capsule administered daily for one month OR 1 placebo patch with patch change every 84 hr for one month in older postmenopausal women
Period: Overall Study
Arm/Group | Young Postmenopausal Women - Estrogen | Older Postmenopausal Women - Estrogen | Young Postmenopausal Women - Placebo | Older Postmenopausal Women - Placebo
Started | 13 | 9 | 8 | 8
Completed | 12 | 9 | 7 | 7
Not Completed | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Younger Postmenopausal Women - Placebo: 1 placebo capsule administered daily for one month OR 1 placebo patch with patch change every 84 hr for one month in younger postmenopausal women
- Total: Total of all reporting groups
Arm/Group | Young Postmenopausal Women - Estrogen | Older Postmenopausal Women - Estrogen | Younger Postmenopausal Women - Placebo | Older Postmenopausal Women - Placebo | Total
Number analyzed (Participants) | 12 | 9 | 7 | 7 | 35
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 51.9 (0.7) | 69.8 (1.1) | 51.1 (1.0) | 71.4 (1.1) | 61.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 7 | 7 | 35
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 9 | 7 | 7 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 0 | 6
  White | 8 | 8 | 5 | 7 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 9 | 7 | 7 | 35

OUTCOME MEASURES:

1. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Changes in Response to Estrogen and Aging - Dorsolateral Pre-frontal Cortex (DLPFC)
Description: Change in extracted beta coefficients of the blood oxygen level dependent (BOLD) signal response to a cognitive task (N-back) in the DLPFC (x,y,z coordinates = -34 44 16) from baseline to 1 month as a function of aging and estrogen (young vs older and estrogen vs placebo). A positive change indicates an increase in oxygen utilization (inferring increased neuronal functioning) between baseline and treatment during the cognitive task, while a negative change indicates a decrease in oxygen utilization between baseline and treatment during the cognitive task.
Time Frame: baseline to 1 month
Population: all young and older postmenopausal women who completed one month of placebo or estrogen and in whom structural and functional MRI data were of significant quality for analysis.
Measure: Mean (Standard Error); unit: linear beta extractions
Groups:
- Young Postmenopausal Women - Placebo; Older Postmenopausal Women - Placebo: 1 placebo capsule administered daily for one month OR 1 transdermal placebo patch with patch change every 84 hr for one month in younger postmenopausal women
Arm/Group | Young Postmenopausal Women - Estrogen | Older Postmenopausal Women - Estrogen | Young Postmenopausal Women - Placebo | Older Postmenopausal Women - Placebo
Number analyzed (Participants) | 12 | 9 | 7 | 7
linear beta extractions | 455.8 (164.3) | -214.4 (90.1) | -348.1 (215.3) | 90.1 (215.3)

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Young Postmenopausal Women - Estrogen: 1 oral capsule (1 mg estradiol) administered daily for one month OR : 1 transdermal estrogen patch (50 mcg/day) with patch change every 84 hr for one month in younger postmenopausal women
- Older Postmenopausal Women - Estrogen: 1 oral capsule (1 mg estradiol) administered daily for one month OR : 1 transdermal estrogen patch (50 mcg/day) with patch change every 84 hr for one month in older postmenopausal women
Arm/Group | Young Postmenopausal Women - Estrogen | Older Postmenopausal Women - Estrogen | Young Postmenopausal Women - Placebo | Older Postmenopausal Women - Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/12 | 2/9 | 1/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Young Postmenopausal Women - Estrogen (N=12) | Older Postmenopausal Women - Estrogen (N=9) | Young Postmenopausal Women - Placebo (N=7) | Older Postmenopausal Women - Placebo (N=7)
anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Experience anxiety in magnet on 1/3 occasions
urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — reported hives 9 days after all study procedures completed
light headed (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Brief period of dizziness one week after completing all procedures. Resolved and no abnormalities noted on clinical MRI.
twisted knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Participant slipped on wet floor after consent and screening but before any study procedures initiated.
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Chronic back condition aggravated during MRI due to positioning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No